CLINICAL TRIAL: NCT03422692
Title: Comparison of Human Amnion Chorionic and Typ1 Bovine Collagen Membranes for Socket Preservation: A Clinical and Histological Study
Brief Title: Socket Preservation: A Clinical and Histological Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Mohanad Al-Sabbagh, Professor and Chief of Periodontology, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Snoasis
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Alveolar Ridge Augmentations
Keywords: Resorbable membrane, amnion-chorion membrane, collagen membrane, ridge preservation.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BioXlude memebrane (Experimental): Subjects in this arm will receive demineralized freeze dried bone allograft covered with BioXclude amnion-chorion membrane following tooth extraction
  Interventions: Biological: BioXclude amnion-chorion membrane
- Mem-Lok (Active Comparator): subjects in this arm will receive demineralized freeze dried bone allograft covered with Mem-Lok collagenous membrane following tooth extraction
  Interventions: Biological: Mem-Lok collagenous membrane

INTERVENTIONS:
Biological: BioXclude amnion-chorion membrane — BioXclude will be used for the prevention of alveolar ridge resorption via socket bone graft and amnion-chorion membrane closure
  Other Names: BioXclude membrane
  Arms: BioXlude memebrane
Biological: Mem-Lok collagenous membrane — Mem-Lok will be used for the prevention of alveolar ridge resorption via socket bone graft and collagenous membrane closure
  Other Names: Mem-Lok
  Arms: Mem-Lok

SUMMARY:
The objective of this study is to investigate the use of human amnion chorion membrane (BioXclude®) as an exposed barrier in ridge preservation and whether the intentional exposure of this membrane to oral environment will adversely affect ridge healing, dimensions, and bone vitality. This is a randomized clinical study.

DETAILED DESCRIPTION:
Alveolar ridge resorption is common sequelae following tooth extraction and presents a challenge for implant placement. The width of the alveolar ridge is known to be resorbed to 30% and 50% of it is original dimension after 3 and 12 months respectively when the extraction socket was left to heal on its own(Schropp, Wenzel et al. 2003). Clinical studies have investigated the socket augmentation technique to prevent the collapse of socket dimension after extraction, and to maintain the ridge width and height for implant placement. This technique includes grafting the socket with bone particulate and then covering the grafted socket with a barrier membrane. (Iasella, Greenwell et al. 2003; Wang and Tsao 2008). In socket augmentation, the role of bone particles is to induce the formation of bone or to provide a scaffold for the new bone formation. The role of the membrane is to keep bone particles within the socket and to exclude the epithelial and connective tissue cells from populating the extraction socket, thus allow the bone cells populating the socket and forming new bone. (Smukler, Landi et al. 1999). The ideal membrane should have no immunological responses, facilitate tissue integration, maintain the clot space, and have good handling properties (Scantlebury 1993; Rakhmatia, Ayukawa et al. 2013). A variety of resorbable and non-resorbable barrier membranes used in socket preservation have been reported in clinical studies. They have clearly shown variable rates of new bone formation prior to implant placement.(Smukler, Landi et al. 1999) (Fotek, Neiva et al. 2009). A xenograft collagen membrane was used in several clinical studies for socket augmentation (Sevor and Meffert 1992; Sevor, Meffert et al. 1993; Iasella, Greenwell et al. 2003; Wang and Tsao 2008).

Another type of resorbable membrane that has been investigated for socket augmentation is the allograft placental membrane. Processed, dehydrated and sterilized human placental amnion chorionic membrane (ACM) has been successfully used in many clinical applications in soft tissue repair and regeneration. (Trelford and Trelford-Sauder 1979; Nakamura, Koizumi et al. 2003).

ACM have also been used in human clinical studies to assess gingival healing and bone formation in augmented sockets and osseous defects.(Wallace 2010; Holtzclaw 2011; Wallace 2011).

In this study, the investigators aim to compare two resorbable membrane (allograft placental-BioXclude versus xenograft collagen- Mem Lok) in order to find out whether one of these membrane could provide better soft tissue healing and better bone quality before implants are placed. Both membranes are FDA approved and tested for human use. Their proposed use in this study is FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* must have an unsalvageable tooth with extraction planned with delayed implant
* extraction sockets must have intact buccal and lingual cortical plates

Exclusion Criteria:

* completely endentulous
* plan for a full mouth tooth extraction
* radiation therapy
* uncontrolled systemic disorders
* acute odontogenic infections
* smoking >10 cigarettes/day
* taking anti-resorptive meds
* pregnant or may become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
bone quality | 19.5 weeks post intervention
  Mean vital bone formation using histomorphometric analysis

SECONDARY OUTCOMES:
Bone quantity | 19.5 weeks post intervention
  vertical and horizontal measurements of alveolar ridge

CONTACTS AND LOCATIONS:
Overall Officials: Mohanad Al-Sabbagh, DDS, MS, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky College of Dentistry, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No